CLINICAL TRIAL: NCT03300258
Title: Robotic Pedaling Therapy for Targeted Neural Plasticity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Original study plan required re-evaluation and the decision was made to pivot to developing tests and exercises on healthy population
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-1279; A196200 (Other: UW Madison); ENGR\MECHANICAL ENGR (Other: UW Madison); Protocol Version 1.8, 3/2017 (Other: UW Madison); 4UL1TR000427-10 (NIH)
Record Dates: First submitted 2017-06-12; First posted 2017-10-03 (Actual); Results first posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Non-Stroke Pilot Group (Other): Robotic therapy. Aerobic therapy. Subjects without stroke, pilot subjects tested during early phases while the device and therapeutic task specifications are developed, and throughout the project while the device and tasks are refined.
  Interventions: Device: Robotic therapy; Device: Aerobic therapy
- Non-Stroke Comparison Group (Other): Robotic therapy. Healthy controls enrolled (age 50-85) to contribute to a normative data set on motor learning using the robotic protocols designed for stroke.
  Interventions: Device: Robotic therapy
- Robotic Training Group (Experimental): Robotic therapy. Subjects with Stroke who will perform the targeted training task: exercise using novel tasks on a robotic recumbent cycle.
  Interventions: Device: Robotic therapy
- Aerobic Training Group (Active Comparator): Aerobic therapy. Subjects with Stroke who will perform aerobic pedaling, duration-matched to the Robotic group.
  Interventions: Device: Aerobic therapy

INTERVENTIONS:
Device: Robotic therapy — The "Robotic" group will use a robotic training protocol to incentivize recovery of motor control by changing task demands throughout the training period. One or more target tasks will be chosen to mimic different sub-functions of gait, including some which are not normally excited in typical cycling behavior. Also, tasks may be designed to target non-gait motions such as hip ab/adduction. The required task may be changed periodically. This therapy protocol will occupy 30 minutes of each training session. Prior to testing, EMG electrodes will be placed on the major muscles of both legs, a procedure that takes roughly 15 minutes. Another 15 minutes is for changing clothes, briefing the subject, and other ancillary study activities. The total time per training session is 1 hour.
  Arms: Non-Stroke Comparison Group; Non-Stroke Pilot Group; Robotic Training Group
Device: Aerobic therapy — The Control group protocol is identical to that of the Robotic group, except the robotically-incentivized exercise is replaced with an aerobic exercise. This intervention emulates a commercial motorized exercise bike to improve cardiovascular unfitness contributions to gait impairment. This therapy implements assist-as-needed and constant-velocity control. The patient's target pedaling speed (e.g. 20 rev/min (to be finalized through pilot tests) and power level (set by heart rate to require approximately 50-70% of maximal oxygen uptake) are set at the beginning of each session and a motor provides assistance or resistance to compensate for the performance of the patient. The exercise will be performed in this mode for 30 minutes per training session.
  Arms: Aerobic Training Group; Non-Stroke Pilot Group

SUMMARY:
The aim of this Pilot study is to determine whether robotically targeted lower-limb pedaling therapy can increase the extent of stroke recovery on behavioral measures and induce brain plasticity as measured by functional magnetic resonance imaging (fMRI). Forty (40) adult stroke patients and 80 healthy controls will be enrolled in this study. Of the 40 patients, half will be randomly assigned to the robotically-targeted training ("robotic") group and will receive training on the targeted training task. The other half of the patients will perform a duration-matched aerobic pedaling exercise ("control" group). All stroke patients will be scanned before and after their training program while performing or imagining simple motor tasks. Behavioral assessments of motor and cognitive capacities will be collected at each timepoint. Healthy control subjects enrolled for device testing (20) will receive up to 5 training sessions in a modified robotic paradigm and 1 fMRI scan, in order to investigate motor learning and brain activity in a novel motor control task. Additional healthy pilot subjects (up to 60) will test training protocols and assessments during preparatory design phases of the project.

ELIGIBILITY:
Patients:

Inclusion criteria:

* Subjects will be stroke patients with persistent moderate unilateral lower extremity deficits, age 50-85 years at time of enrollment.
* Time since stroke will be greater than 6 months ("chronic" stroke survivors).
* Persistent moderate unilateral lower-limb impairment (defined as NIH Stroke Scale - Motor Leg section score of 1-2, to be discussed with the patient verbally during phone screening and assessed by the investigator during the initial enrollment visit).
* Fluent in spoken and written English

Exclusion criteria:

* Allergy to electrode gel, surgical tape and metals.
* Subjects under treatment for infectious diseases will be excluded from the study.
* Women who are pregnant or planning to become pregnant during the course of the study will be excluded.
* Contraindications for MRI
* Age over 85 years at time of enrollment.

Healthy Controls:

Inclusion criteria:

* Ages 18-85 years
* Non-Stroke Group 1 ("Matched Controls"): 50-85 years old at time of enrollment, to match the population of stroke patients to be studied
* Non-Stroke Group 2 ("Pilot Controls"): 18-50 years old at time of enrollment (Pilot subjects to be initially enrolled early in the design phase of the study, and with enrollment ongoing throughout the study to continue development.)
* No known neurologic, psychiatric or developmental disability.
* Fluent in spoken and written English

Exclusion criteria:

* Allergy to electrode gel, surgical tape, and metals.
* Subjects under treatment for infectious diseases will be excluded from the study.
* Women who are pregnant or planning to become pregnant during the course of the study will be excluded.
* Contraindications for MRI
* Age over 85 years at time of enrollment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter G Adamczyk, Ph.D., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy participants were recruited from June 2019 to June 2022.
Pre-assignment Details: Original study plan required re-evaluation and the decision was made to pivot to developing tests and exercises on healthy population. A clinical trial was not conducted.
Groups:
- Non-Stroke Pilot Group: Robotic therapy and Aerobic therapy
  Subjects without stroke, pilot subjects tested during early phases while the device and therapeutic task specifications are developed, and throughout the project while the device and tasks are refined.
- Non-Stroke Comparison Group: Robotic therapy
  Healthy controls enrolled (age 50-85) to contribute to a normative data set on motor learning using the robotic protocols designed for stroke.
- Robotic Training Group: Robotic therapy
  Subjects with Stroke who will perform the targeted training task: exercise using novel tasks on a robotic recumbent cycle.
Period: Overall Study
Arm/Group | Non-Stroke Pilot Group | Non-Stroke Comparison Group | Robotic Training Group | Aerobic Training Group
Started | 44 | 0 | 0 | 0
Group 1: Reaching Against a Spring-Like Torque | 12 | 0 | 0 | 0
Group 2: Reaching Against a Damper-like Force | 11 | 0 | 0 | 0
Group 3: Half-Reversed Cycling Task | 21 | 0 | 0 | 0
Completed | 44 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Non-Stroke Pilot Group
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 25
  More than one race | 11
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Change in Six Minute Walk Test (6MWT) Distance
Description: A simple series of laps along a 30 m straight path in a level hallway.
Time Frame: Baseline and at 5 weeks
Population: Healthy Pilot Group participants were enrolled and the study team learned that the protocol was insufficient to test the hypothesis. No data were collected for this measure.
Arm/Group | Non-Stroke Pilot Group | Non-Stroke Comparison Group | Robotic Training Group | Aerobic Training Group
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Change in Brain Activity in and Near Affected Areas, Through Functional MRI (fMRI)
Description: fMRI scans will be used to measure task-specific cortical activity in sensorimotor areas during physical stepping with an MRI-compatible stepping machine, or imagined/visualized cycling.
Time Frame: Baseline and at 5 weeks
Population: as for outcome 1
Arm/Group | Non-Stroke Pilot Group | Non-Stroke Comparison Group | Robotic Training Group | Aerobic Training Group
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Change in Timed Up-and-Go Test (TUG)
Description: A simple timed test of how long it takes to stand up, walk 10 feet, turn around, return to the starting point, and sit down.
Time Frame: Baseline and at 5 weeks
Population: as for outcome 1
Arm/Group | Non-Stroke Pilot Group | Non-Stroke Comparison Group | Robotic Training Group | Aerobic Training Group
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Change in Self-Selected Walking Speed (SSWS)
Description: A simple test of the speed a person chooses to walk over a 5-meter distance
Time Frame: Baseline and at 5 weeks
Population: as for outcome 1
Arm/Group | Non-Stroke Pilot Group | Non-Stroke Comparison Group | Robotic Training Group | Aerobic Training Group
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Change in Fastest Comfortable Walking Speed (FCWS)
Description: A similar test of the "fastest comfortable speed" a person can use to walk over the 5-meter distance
Time Frame: Baseline and at 5 weeks
Population: as for outcome 1
Arm/Group | Non-Stroke Pilot Group | Non-Stroke Comparison Group | Robotic Training Group | Aerobic Training Group
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Change in Center of Pressure (COP) Characteristics
Description: Movement of the Center of Pressure during standing, with eyes open and eyes closed. With eyes open, subjects focus their eyes on a spot on the wall in front of them. Metrics of COP control include excursion, average velocity, standard deviation, and an estimate of center of mass location.
Time Frame: Baseline and at 5 weeks
Population: as for outcome 1
Arm/Group | Non-Stroke Pilot Group | Non-Stroke Comparison Group | Robotic Training Group | Aerobic Training Group
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Post Hoc Outcome: Reaction Time in "Medium" Catch Trials
Description: The test involved reaching against spring-like torque, where the spring stiffness was mostly constant but was changed unexpectedly by the computer in different trials. Reaction time definition: time from a visual and auditory cue to initial movement.
  Participants were "Trained" with mostly a Low or High stiffness (each in a separate block of reaches) and had "Catch" trials when the stiffness was changed to Medium.
  "Low" stiffness = 10 Newton meter per radian (Nm/rad); "Medium" stiffness = 20 Nm/rad; "High" stiffness = 30 Nm/rad
Time Frame: 1 visit roughly 3 hours
Population: Original study plan required re-evaluation and the decision was made to pivot to developing tests and exercises on healthy population. A clinical trial was not conducted. Summary Data collected from experimental tasks in development are reported here as post-hoc outcomes.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Group 1: Reaching against a Spring-Like Torque experiment
Arm/Group | Group 1
Number analyzed (Participants) | 12
seconds
  Train High, Catch Medium | 0.366 (0.038)
  Train Low, Catch Medium | 0.375 (0.037)

8. Post Hoc Outcome: Movement Settling Time: Reaching Against a Spring-Like Torque
Description: The test involved reaching against spring-like torque, where the spring stiffness was mostly constant but was changed unexpectedly by the computer in different trials. Movement Settling Time definition: time for crank angle to settle between 40 and 50 degrees, when the central target was 45 degrees.
  "Low" stiffness = 10 Nm/rad; "Medium" stiffness = 20 Nm/rad; "High" stiffness = 30 Nm/rad
  "Catch trials" are unexpected medium stiffness setting, unpredictably spaced.
Time Frame: 1 visit roughly 3 hours
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Group 1
Number analyzed (Participants) | 12
seconds
  "high" stiffness training | 1.21 (0.068)
  "low" stiffness training | 1.24 (0.071)
  "catch medium" trials when training was "high" | 1.29 (0.079)
  "catch medium" trials when training was "low" | 1.40 (0.096)

9. Post Hoc Outcome: Undershoot and Overshoot in Catch Trials
Description: The test involved reaching against spring-like torque, where the spring stiffness was mostly constant but was changed unexpectedly by the computer in different trials. All participants had a block with "Low" training, called "Train Low Catch Medium", and a separate block with "High" training, called "Train High Catch Medium".
  Undershoot: initial reach showed undershoot relative to the target crank angle of 45 degrees, with the value measured as the local minimum as the pedal momentarily stopped and went backward.
  Overshoot: initial reach showed overshoot beyond the target crank angle of 45 degrees, with the value measured as the maximum angle during that period.
Time Frame: 1 visit roughly 3 hours
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Group 1
Number analyzed (Participants) | 12
degrees
  Undershoot | 37.3 (2.1)
  Overshoot | 52.4 (2.6)

10. Post Hoc Outcome: Movement Settling Time: Reaching Against a Damper-Like Force
Description: The test involved reaching against viscous damper torque, where the damping constant (units: Nm/(rad/s) = torque produced by the robot per rad/s of crank velocity) was changed by the computer in a structured but unpredictable sequence, across the trials. Movement settling time is defined as time for crank angle to settle between 40 and 50 degrees, when the central target was 45 degrees.
  Low damping = 3 Nm/(rad/s), High damping = 9 Nm/(rad/s).
Time Frame: 1 visit roughly 3 hours
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Group 2: Reaching against a damper-like force experiment
Arm/Group | Group 2
Number analyzed (Participants) | 11
seconds
  high damping | 1.21 (0.040)
  low damping | 1.17 (0.056)

11. Post Hoc Outcome: Movement Settling Time With Damping Level Cued Visually
Description: The test involved reaching against viscous damper torque, where the damping constant (units: Nm/(rad/s) = torque produced by the robot per rad/s of crank velocity) was changed by the computer in a structured but unpredictable sequence, across the trials. Movement settling time is defined as time for crank angle to settle between 40 and 50 degrees, when the central target was 45 degrees. In this experiment, the damping level was visually cued. Low damping = 3 Nm/(rad/s), High damping = 9 Nm/(rad/s)
Time Frame: 1 visit roughly 3 hours
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Group 2
Number analyzed (Participants) | 11
seconds
  High Damping Cued Visually | 1.16 (0.041)
  Low Damping Cued Visually | 1.13 (0.030)

12. Post Hoc Outcome: Number of Participants Who Completed the Half-Reversed Cycling Task
Description: The effect of pushing on one specific pedal was reversed by the computer in its calculation of how to move the crank; the other pedal had a physically typical effect. The task was to cause this complex system to move the crank at a constant 20 RPM forward speed (i.e., minimize the error in speed from this target). Reported here are the number of participants who completed this task.
Time Frame: Five training sessions of 45 minutes, each on a different day within roughly one week. Additionally, a 6th session with the effects of the two pedals switched
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Groups:
- Group 3: Half-Reversed Cycling Task
Arm/Group | Group 3
Number analyzed (Participants) | 21
Participants | 21

ADVERSE EVENTS:
Time Frame: up to 1 week
Arm/Group | Non-Stroke Pilot Group
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 0/44

LIMITATIONS AND CAVEATS:
Original study plan required re-evaluation and the decision was made to pivot to developing tests and exercises on healthy population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT03300258/Prot_SAP_000.pdf